CLINICAL TRIAL: NCT02027298
Title: Abatacept for Patients With Inflammatory Arthritis Associated With Sjögren's Syndrome: an Open-Label Phase II Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Enrollment
Sponsor: The Cleveland Clinic (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-Yao-2012001
Record Dates: First submitted 2013-11-18; First posted 2014-01-06 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2015-02

CONDITIONS: Primary Sjogren's Syndrome; Secondary Sjogren's Syndrome; Inflammatory Arthritis; Rheumatoid Arthritis
Keywords: Abatacept; Sjogren's Syndrome; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Sjogren's Syndrome | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abatacept (Experimental): Abatacept by SC injection of 125 mg weekly for 6 months
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — by SC injection of 125 mg weekly for 6 months
  Other Names: Orencia

SUMMARY:
The primary purpose of this pilot study is to evaluate the efficacy and safety of Abatacept in subjects with Sjogren's Syndrome (SS). This clinical trial study will enroll and treat 15 subjects with active moderate and severe inflammatory arthritis associated with primary Sjogren's syndrome (pSS) and secondary Sjogren's sybdrine (sSS) with Rheumatoid Arthrits (RA). All subjects will receive Abatacept weekly by Subcutaneous (SC) dosing. Subjects will receive Abatacept by SC injection of 125 mg on day 1 and followed by 125 mg SC weekly thereafter.

DETAILED DESCRIPTION:
Sjogren's Syndrome (SS) is a common systemic autoimmune disease, including primary and secondary form. About 30% of RA are associated with sSS (1) Tumor necrosis factor alpha inhibitors (TNFa-Is) have been tried in this population without success. Abatacept (CTLA4-Ig) is comprised of the ligand-binding domain of CTLA4 plus human immunoglobulin and represents a novel therapeutic costimulation blocker that modulates the signal required for full T cell activation. Studies have shown that activated CD4 T cells play a role in the pathogenesis of SS, indicating Abatacept might be a useful therapeutic intervention in SS. Subjects who are receiving non-biologic immunosuppressive medications consisting of hydroxychloroquine, methotrexate (MTX), sulfasalazine, or leflunomide, at the time of enrollment will remain on these medications without dosage alteration. Efficacy and Safety data will be collected at the time of each clinic visit. The treatment closing date will occur 6 months after enrollment of each subject. Subjects will be followed at 1, 2, 3, 4, 5, and 6 months. Laboratory studies associated with the clinical trial will test potential autoantibody production for systemic autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Sjogren's Syndrome
2. Patients are at least 18 years or older
3. Patients should have either pSS and/or sSS associated with RA, and must have active moderate to severe inflammatory arthritis as defined by painful joint counts (≥5) and swollen joint counts (≥5), or DAS28 scores>3.2.
4. One non-biologic DMARD will be permitted.
5. These patients will be willing and able to comply with treatment and follow-up procedures.
6. These patients will be willing and able to provide written informed consent.
7. Both women and men of child bearing age must be willing to use an effective means of birth control while receiving treatment throughout participation in this study. Effective contraception methods include abstinence, oral contraceptives (birth control pills), IUD, diaphragm, Norplant, approved hormone injections, condoms, or medical sterilization.

Exclusion Criteria:

1. Patients will be excluded if they have a concomitant disorder requiring systemic glucocorticoid (GC) therapy (prednisone >10 mg daily or GC equivalent), have organ-threatening features, and have any investigational drug including biologics within 28 days of study entry.
2. History of cancer or diabetes mellitus
3. Use of tricyclic antidepressants or anticholinergics
4. Evidence of active infection or chronic infection including human immunodeficiency virus (HIV), tuberculosis (TB), hepatitis C, or a positive hepatitis B surface antigen.
5. Patients with latent TB if not treated with isoniazid for at least 4 weeks prior to receiving the study drug
6. Radiographic evidence of COPD, emphysema, and/or interstitial lung disease.
7. Subjects who are pregnant or who are nursing infants
8. Patients with cytopenia: platelet count <80,000/mm3, absolute neutrophil count<1500/mm3, hematocrit < 20%.
9. Patients with renal insufficiency defined by a serum creatinine of greater than or equal to 2.0 mg/dL or creatinine clearance of less than or equal to 35 ml/min.
10. Use of illegal drugs.
11. A live vaccination fewer than 4 weeks before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of Abatacept in patients with inflammatory arthritis and Sjogren's Syndrome | 6 months
  To determine the efficacy for inflammatory arthritis of Abatacept in patients with both pSS and sSS. The primary efficacy endpoint for determining the efficacy is the proportion of patients meeting the ACR 20% improvement criteria at month 6.

SECONDARY OUTCOMES:
Increase or change in autoantibody profile | Month 3, 6 and 3 month follow up
  A secondary endpoint is to assess autoantibody production as measured by Bioplex2200, including antinuclear antibodies (ANA), anti-ENA (Sm, RNP, SSA, SSB, chromatin, Scl70 and centromere) antibodies, anti-dsDNA antibodies, Complement 3 (C3)/Complement 4 (C4), immunoglobulin (Ig), erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP).
Explore the potential efficacy of Abatacept in the exocrine glandular function | Month 1, 3 and 6
  The last efficacy endpoint is to explore the efficacy of Abatacept in the exocrine glandular function including assessment of xerophthalmia and xerostomia using 0-100 mm visual analog scale (VAS)(29) and functional measurement of salivary gland and lacrimal gland.

CONTACTS AND LOCATIONS:
Overall Officials: Qingping Yao, MD, Ph.D, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States